CLINICAL TRIAL: NCT04542200
Title: Workforce Serosurveillance to Track Long-term Modifications to COVID-19 Exposure Due to Factors in the Built Environment
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0668
Record Dates: First submitted 2020-09-08; First posted 2020-09-09 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Antibody testing — The antibody results include understanding modifications from environments at work and the community.

SUMMARY:
The goal, with this study, is to leverage Northwell Health System's diverse workforce and robust testing structures, to contribute data-driven, evidence-based strategies to better understand the sustained prevalence of antibodies and how conferred immunity may be modified by environmental factors. The objective is to investigate the COVID-19/SARS-CoV-2 disease prevalence and trajectory over time, by conducting follow-up antibody testing on employees who consented to participate in research during the initial workforce offering. From 70,812 employees contacted, 46,117 were tested and received initial results. Of those participants, approximately, 32,000 agreed to be re-contacted, and 34,000 consented to research. The investigators plan to conduct an additional five rounds of testing that would sample individuals over a two-year period. This study is significant because it leverages Northwell Health's advanced laboratory systems to conduct serosurveillance of antibodies to COVID-19/SARS-CoV-2 across a large and diverse workforce, while taking into account the contextual environmental and occupational exposures that may modify continued immunity to the virus. Northwell Health's employee health services (EHS) is poised to act quickly to adapt policies and practices, where needed, to protect the workforce. The study is also innovative because it will be linking work environment and community measures with COVID-19 seropositive prevalence patterns over time, to build a better understanding of the disease and its controls at the population level. The expected outcomes include serial serology results as a measure of full or partial short-term (6 months) and long-term (2 year) immunity to re-infection and recognition of local environmental factors (e.g., building ventilation rates, zip code, air quality indicators) that could modify this immunity and assist with protecting the workforce and surrounding community. These results could inform national and global policies.

DETAILED DESCRIPTION:
The objective of this study is to understand the COVID-19/SARS-CoV-2 disease incidence, prevalence, and trajectory over time, by conducting follow-up antibody testing on employees by first following up with the approximately 5,600 team members who were positive and then extending the invitation to the remaining team members (approximately 65,212).

Aim 1) Follow those who tested positive during prior institutional antibody testing to better understand whether IgG or total antibody measures confer continued immunity; hypothesis 1 is that prior infection will be protective and that restricting testing to prior positives, reduces impact of false positive results due to low prevalence populations. Over a 1.5 year period, testing will be repeated on seropositive individuals in January 2021, May 2021, September of 2021, January 2022, and May 2022.

The results will be to document antibody seropositivity and continued presence of immunity over time. The study investigators will invite those positive Northwell team members to participate in a research study that has the aim of testing for continued presence of antibodies to COVID-19, to understand trends over time.

Aim 2) Continue to document seroconversion rates and distribution of exposure to COVID-19 across the entire remaining workforce; hypothesis 2 is that employees will have lower rates than the general population, even though false positive serology results will be highly dependent upon New York State positive prevalence rates. Over the same 1.5 year period as in Aim 1, testing will be repeated for all workforce participants who previously tested negative and others interested in participating for the first time in May 2021 (or September 2021) and May 2022.

Aim 3) Track any associations between engineering, administrative, and personal protective equipment (PPE) policies across the health system and whether these continue to be protective and adapt to disease/viral behavior over time; hypothesis 3 is that Northwell Health policies are proactive and protective and that co-exposures to environmental factors in the workplace and community are measurable and remediable with respect to their effects on COVID-19 infection rates. The investigators propose to complete three things. First, they will be linking job title, department, and industry codes from participant records, with occupational indices of workplace exposure, such as O*Net. This will create a job or task exposure matrix (JEM) for job groups in the Northwell Health system. This JEM will reflect conventional understanding of job level exposure risk estimates to work stressors that may be physical (e.g., heavy loads), psychosocial (e.g., job demand/control), noise, and chemical (e.g., peracetic acid cleaners). Second, they will link departmental level policy information on personal protective equipment (PPE) for each job/task; administrative policies on work hours for the job and chemicals used for infection control at the unit level; and engineering (ventilation rates) at the building and unit level (e.g., air changes per hour and occupancy limits). This institutional policy information will be gathered from January 2021 to each wave of data collection. Any changes in policy will be documented and the most recent policy will be linked with the job title information. Third, the investigators will integrate community variable census information (at the census tract or zip code level) on neighborhood air quality, poverty rates, language predominance, nativity (US or other), and household density. The study will include travel distance to work and transportation mode.

The investigators anticipate that findings from this work, particularly from Aim 3, have implications that extend to communities across New York State (Northwell Health is the largest employer in New York and its employee residences and work locations span every county). They also believe that this work has broader national and international relevance, as the world continues global efforts to navigate a built environment in which SARS-CoV-2 now exists in a pandemic. The strengths of this study are that it accesses a large population sample of 70,812 people that is diverse and also self-contained, whereby, multiple work, home, and environmental factors can be measured alongside trajectories in COVID-19 prevalence. The population is economically and culturally diverse, even by global standards, and includes Queens County that has recorded some of the highest seropositivity rates to date.

ELIGIBILITY:
Inclusion Criteria:

* Northwell Health employees

Exclusion Criteria:

* Those not employed at Northwell Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Working population of Northwell Health
Sampling Method: Non-Probability Sample
Enrollment: 40132 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 antibodies | Two years
  serology testing

CONTACTS AND LOCATIONS:
Overall Officials: Grace Sembajwe, ScD, Principal Investigator — Feinstein Institutes for Medical Research, Northwell Health
Locations (1):
- Feinstein Institutes for Medical Research, Northwell Health, Great Neck, New York, United States